CLINICAL TRIAL: NCT06655545
Title: A Single-center, Real-world Study Exploring the Guidance of FES-PET for First-line Treatment of HR Positive, HER2 Negative Unresectable or Metastatic Breast Cancer Patients
Brief Title: 18F-fluoroestradiol (18F-FES) PET/CT Guided First-line Treatment for HR+/HER2- Metastatic Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-31
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: chemotherapy; CDK4/6 inhibitors; 18F-fluoroestradiol (18F-FES) PET/CT; HR positive; HER2 negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- FES-guided CDK4/6 inhibitor plus endocrine therapy cohort: The group guided with FES-PET using a CDK4/6 inhibitor plus ET.
- FES-guided chemotherapy cohort: The group guided with FES-PET using chemotherapy.
- Non-FES-guided CDK4/6 inhibitor plus endocrine therapy cohort: The group examined without FES-PET using a CDK4/6 inhibitor plus ET.
- Non-FES-guided chemotherapy cohort: The group examined without FES-PET using chemotherapy.

SUMMARY:
A single-center, real world study to evaluate the role of FES-PET in guiding the first-line treatment of HR+/HER2- MBC patients.

ELIGIBILITY:
Inclusion Criteria:

1. age >= 18 years old;
2. Patients who were diagnosed as HR Positive, HER2 Negative recurrent unresectable (local or regional) or stage IV (M1) breast cancer between January 2020 to February 2024;
3. Received CDK4/6 inhibitor plus endocrine treatment or chemotherapy as first-line therapy for at least one cycle;
4. Complete medical history was available.

Exclusion Criteria:

1. Medical history was incomplete.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as HR Positive, HER2 Negative recurrent unresectable (local or regional) or stage IV (M1) breast cancer between January 2020 to February 2024.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  progression-free survival

SECONDARY OUTCOMES:
OS | 6 weeks
  overall-survival

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China